CLINICAL TRIAL: NCT02290262
Title: SheppheartCABG. A Randomised Clinical Trial of a Comprehensive Physical and Psycho-educative Rehabilitation Programme Plus Usual Care Versus Usual Care in Phase 1 Rehabilitation After Coronary Artery Bypass Grafting
Brief Title: SheppHeartCABG - Phase One Rehabilitation After Coronary Artery Bypass Grafting
Acronym: SheppHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Senior researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SheppHeartCABG RCT
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Ischaemic Heart Disease
Keywords: Heart disease; Phase one rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive phase one rehabilitation (Experimental): Patients allocated to the experimental group receive a rehabilitation programme consisting of physical exercise and psycho-education plus usual care.
  Interventions: Other: Comprehensive phase one rehabilitation
- Usual care (No Intervention): The control group will receive usual care alone.

INTERVENTIONS:
Other: Comprehensive phase one rehabilitation — Patients allocated to the experimental group receive a rehabilitation programme consisting of physical exercise and psycho-education.
  The physical exercises consist of; breathing exercises with and without using incentive spirometry with expiratory positive pressure airway, walking and cycling exercises and neck/shoulder exercises during hospitalisation and an exercise programme running from discharge until 4 weeks following surgery. The psycho-educative rehabilitation programme consists of four psycho-educative consultations with a specially trained nurse.
  Arms: Comprehensive phase one rehabilitation

SUMMARY:
Background: Patients undergoing coronary artery bypass graft surgery often experience a range of problems and symptoms related to the procedure and the underlying heart disease.These problems include anxiety and depressive symptoms, immobility issues, complications such as wound seeping, neck and shoulder pains, interrupted and insufficient sleep. No studies have tested a combined intervention on phase 1 rehabilitation in coronary artery bypass graft surgery patients. However, randomised trials with either a physical or a mental part have been conducted with positive result, but evidence is lacking for a combined intervention. Before a large randomised trial was set up a pilot trial was conducted to evaluate the feasibility of patient recruitment and intervention: to test the safety and tolerability of the intervention by patients and to provide outcome data for sample size calculations. The SheppHeartCABG pilot showed trial feasibility, safety and sufficient inclusion rate and high compliance with most elements. Outcome data from the pilot trial has been used to sample size and power calculation in this randomised clinical trial.

Objective: The objective of this trial is to investigate the benefits and harms of a phase 1 comprehensive cardiac rehabilitation programme consisting of an exercise-training and a psycho-educative component, including plus treatment as usual in patients who undergo coronary artery bypass grafting.

DETAILED DESCRIPTION:
Background: Patients undergoing coronary artery bypass grafting surgery often experience a range of problems and symptoms related to the procedure and the underlying heart disease. These problems include anxiety and depressive symptoms, immobility issues, complications such as wound seeping, neck and shoulder pains, interrupted and insufficient sleep. Over the last 2 decades, cardiac rehabilitation has become recognized as a significant component in the continuum of care for persons with cardiovascular disease. Furthermore, cardiac rehabilitation has undergone a significant evolution moving from a focused exercise intervention to a comprehensive disease management program. In Guidelines for Coronary Artery Bypass Graft Surgery cardiac rehabilitation is described as including early ambulation during hospitalisation and outpatient prescriptive exercise training beginning 6-8 weeks following surgery. Our hypothesis is that a comprehensive rehabilitation programme including physical exercise with moderate intensity and a psycho-educative component can begin in the early postoperative phase during hospitalising.

No studies have tested a combined intervention on phase 1 rehabilitation in coronary artery bypass graft surgery patients. However, randomised trials with either a physical or a mental part have been conducted with positive result, but evidence is lacking for a combined intervention. Before a large randomised trial was set up a pilot trial was conducted to evaluate the feasibility of patient recruitment and intervention: to test the safety and tolerability of the intervention by patients and to provide outcome data for sample size calculations. The SheppHeartCABG pilot showed trial feasibility, safety and sufficient inclusion rate and high compliance with most elements. Outcome data from the pilot trial has been used to sample size and power calculation in this randomised clinical trial.

Objective: The objective of this trial is to investigate the benefits and harms of a phase 1 comprehensive cardiac rehabilitation programme consisting of an exercise-training and a psycho-educative component, including plus treatment as usual in patients who undergo coronary artery bypass grafting.

Design: SheppHeartCABG is an investigator-initiated randomised clinical trial with 1:1 randomisation from two sites to a comprehensive physical and psycho-educative rehabilitation programme plus usual care or usual care alone, with blinded outcome assessment.

Population: Patients 18 years or older with ischaemic heart disease, who have to undergo elective coronary artery bypass grafting, who speak and understand Danish and who provide a written informed consent will be included. The following patients will be excluded from the trial: patients at intermediate or high risk to their cardiovascular status according to guidelines, patients with neurological or orthopaedic deficits which prevent training and patients who do not wish to participate.

Number of participants: 326 participants will be included.

Interventions: All patients - both in the intervention group and in the control group - receive usual care. Patients allocated to the experimental group receive a rehabilitation programme consisting of physical exercise and psycho-education. The control group will receive usual care alone. The physical exercises consist of; breathing exercises with and without using incentive spirometry with expiratory positive pressure airway, walking and cycling exercises and neck/shoulder exercises during hospitalisation and an exercise programme running from discharge until 4 weeks following surgery. The psycho-educative rehabilitation programme consists of four psycho-educative consultations with a specially trained nurse. The last consultation will take place 4 weeks following surgery.

Outcomes: Primary outcome is physical capacity measured by 6-minute walk test 4 weeks following surgery. Secondary outcomes; perceived mental and physical(SF 12), health-related quality of life (HeartQoL), anxiety and depression (HADS), sleep (PSQI), pain (ÖMPSQ) and leg endurance and strength (sit and stand test). Explorative outcomes are; fatigue (MFI-20), physical activity (IPAQ), cognitive and emotional representation of illness (B-IPQ) and self-rated health (EQ-5D).

Safety: There are no previous reports of risks associated with psycho-educational consultations. Physical exercise is tested extensively in patients with heart disease and is considered safe and will meet the applicable requirements for safety during training of cardiac patients. The interventions are considered safe for patients at low risk according to their cardiovascular status.

Ethical considerations: The trial is performed in accordance with the Declaration of Helsinki in its latest form. All patients must give informed consent prior to participation and the trial is initiated after approval by the Danish Data Protection Agency and the regional ethics committee. The trial will be registered at www.clinicalTrials.gov before randomisation of the first participant.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with ischaemic heart disease,
* Who have to undergo elective coronary artery bypass grafting,
* Who speak and understand Danish and
* Who provide a written informed consent will be included.

Exclusion Criteria:

Patients will be excluded from the trial:

* Patients at intermediate or high risk to their cardiovascular status according to guidelines,
* Patients with neurological or orthopaedic deficits which prevent training and
* Patients who do not wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 4 week
  Primary outcome is physical capacity measured by 6-minute walk test 4 weeks following surgery.

SECONDARY OUTCOMES:
Composite secondary outcomes | 4 week
  . Secondary outcomes consists of perceived mental and physical(SF 12), health-related quality of life (HeartQoL), anxiety and depression (HADS), sleep (PSQI), pain (ÖMPSQ) and leg endurance and strength (sit and stand test) measured 4 weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Selina Berg, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Hjertecentret, Copenhagen University Hospital, Rigshospitalet, Blegdamsvej 9, Copenhagen, OE, Denmark

REFERENCES:
- [Derived] Hojskov IE, Moons P, Hansen NV, La Cour S, Olsen PS, Gluud C, Winkel P, Lindschou J, Thygesen LC, Egerod I, Berg SK. SheppHeartCABG trial-comprehensive early rehabilitation after coronary artery bypass grafting: a protocol for a randomised clinical trial. BMJ Open. 2017 Jan 17;7(1):e013038. doi: 10.1136/bmjopen-2016-013038. PMID 28096255